CLINICAL TRIAL: NCT03875378
Title: Transdermal Estrogen for the Treatment of Bone Loss in Women With Anorexia Nervosa
Brief Title: Transdermal Estrogen in Women With Anorexia Nervosa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pouneh K. Fazeli, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Pouneh K. Fazeli, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19070395; R01HD099139 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: Bone mineral density; Estrogen
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdermal estrogen/progesterone (Experimental): Transdermal estradiol (0.045mg)/levonorgestrel (0.015mg) patch applied weekly for 18 months
  Interventions: Drug: Transdermal estrogen
- Placebo (Placebo Comparator): Placebo patch applied weekly for 18 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Transdermal estrogen — Transdermal estradiol (0.045mg)/levonorgestrel (0.015mg) weekly patch
  Arms: Transdermal estrogen/progesterone
Drug: Placebos — Placebo weekly patch
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled study investigating the use of physiologic, transdermal estrogen for low bone mass in adult women with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa is a prevalent psychiatric with a lifetime prevalence of up to 2.2%. Among the many medical co-morbidities associated with anorexia nervosa, the most common is significant bone loss, which can persist despite weight recovery. Nearly 90% of women with anorexia nervosa have osteopenia and this low bone mass is associated with an increased fracture risk. Nearly 30% of women with anorexia nervosa report a history of a fracture and a prospective study demonstrated a 7-fold increased risk of fracture in women with anorexia nervosa compared to age-matched controls. Because anorexia nervosa is a chronic disease that can persist despite psychiatric and nutritional counseling, the bone loss and increased fracture risk can persist and lead to lifelong morbidity. Therefore, finding a treatment for bone loss associated with anorexia nervosa is of critical importance.

This 18-month randomized, placebo-controlled study will investigate in women (ages 20 to 45 years old) with anorexia nervosa whether treatment with transdermal estrogen replacement will increase bone mineral density (BMD).

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 19-45 years of age
3. DSM-5 psychiatric criteria for anorexia nervosa
4. <85% of ideal body weight as defined by the 1983 Metropolitan Life Insurance Height and Weight Tables
5. Amenorrhea
6. T-score of < -1.0 at spine or hip

Exclusion Criteria:

1. Diseases known to affect bone metabolism, including untreated thyroid dysfunction, vitamin D deficiency, Cushing's syndrome, diabetes mellitus or renal insufficiency (eGFR < 60)
2. Personal history of venous or arterial clot
3. History of stroke or myocardial infarction
4. History of hypercoagulable disorder
5. Personal history or history of a first-degree relative with breast cancer
6. History of hereditary angioedema
7. Any medication known to affect bone metabolism, including systemic glucocorticoids within three months of the baseline visit, depot medroxyprogesterone within 6 months of the baseline visit, oral bisphosphonates within one year of the baseline visit or IV bisphosphonates within three years of the baseline visit
8. Bone fracture within the prior 12 months
9. Serum potassium < 3.0 meq/L, serum ALT > 3 times the upper limit of normal or Hemoglobin < 10 g/dL
10. Fasting serum triglyceride level > 150 mg/dL
11. Pregnant or breastfeeding (or desiring pregnancy within the next 18 months)
12. Active substance abuse
13. Elevated PTH level
14. 25-OH vitamin D level < 20 ng/mL
15. Low phosphorus level

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density at 18 months | Baseline, 18 months
  Change in lumbar spine bone mineral density at 18 months

SECONDARY OUTCOMES:
Change in bone mineral density at hip at 18 months | Baseline, 18 months
  Change in total hip bone mineral density at 18 months
Change in bone mineral density at femoral neck at 18 months | Baseline, 18 months
  Change in femoral neck bone mineral density at 18 months
Change in parameters of bone microarchitecture at 18 months | Baseline, 18 months
  Change in microarchitectural parameters as measured by high-resolution peripheral quantitative CT at 18 months
Change in estimated bone strength at 18 months | Baseline, 18 months
  Change in estimated bone strength as assessed by finite element analysis at 18 months
Change in vertebral fractures at 18 months | Baseline, 18 months
  Change in vertebral fractures as assessed by vertebral fracture assessment at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pouneh Fazeli, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and behavioral data from interviews with the subjects, laboratory data from blood specimens provided and radiologic images of subjects with anorexia nervosa. Because anorexia nervosa is a psychiatric disease and we will be collecting identifying information, even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that the information disclosed by the subjects should be protected in the most stringent way possible in order to prevent possible identification of subjects. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after publication and no pre-specified end date.